CLINICAL TRIAL: NCT03578679
Title: Study of the Therapeutic Efficacy of the Combination Azithromycin + Ivermectin in the Treatment of Pediculosis in Senegal (IVERAZITH)
Brief Title: Treatment of Pediculosis (Head Lice) in Senegal
Acronym: IVERAZITH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEN17/16
Record Dates: First submitted 2018-06-21; First posted 2018-07-06 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-07

CONDITIONS: Pediculoses
MeSH Terms: conditions — Lice Infestations | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Interventional prospective study with only one arm
Masking Description: Evaluation of therapeutic efficacy of a combination of two usual drugs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HEGOR/AZICUR shampoo solution (Experimental): At D1, shampoo AZICUR liquid formulation in infested persons aged 0 to 6 years and / or less than 15 kg, also apply the combination HEGOR / AZICUR solution shampoo in women pregnant or lactating women not eligible for treatment with Ivermectin, to prevent them from contaminate treated participants who are very close to them or share the same bed or same bench table at school.
  Interventions: Drug: Ivermectin Oral Product

INTERVENTIONS:
Drug: Ivermectin Oral Product — treatment of pediculosis (head lice)
  Other Names: Azithromycine oral Product

SUMMARY:
This is a prospective single-arm interventional study evaluating Therapeutic efficacy of a combination of two pharmaceutical drugs, Azithromycin (AZIT) and Ivermectin (IVER) administered orally in the treatment of head lice infestations. In case of persistence of lice and / or nits on day 7, a second oral administration of combination Azithromycin + Ivermectin will be considered.

The duration of the study period is 4 months, ie 1 month and ½ of inclusion and 2 months and ½ feedback. There will be a site initiation visit "site initiation visit" before inclusions at D-7, two monitoring visits and a closing visit "close out visit" at the end of the follow-up at 4 months.

DETAILED DESCRIPTION:
The investigators will perform a clinical trial of efficacy, single-arm, until D28 from volunteer subjects infested with head lice.

The two villages of the study (Dielmo and Ndiop) will be visited to explain the protocol and obtain community permission to work on it. Schools will also be visited to inform teachers and explain the protocol. The search for lice will be done by village women recruited for this purpose. A systematic census by family will be performed. A clinical examination of the hair will detect the persons infested with lice. On D-1, individual informed consent (an assent for participants between the ages of 15 and 18) will be systematically obtained before inclusion.

At D1, an interview and a complete clinical examination will be done on each subject consenting. All volunteers meeting the inclusion criteria will be taken on a single arms. For each voluntary participant selected fasting 1 hour before, the treatments will be administered by the investigators of the study. After taking the AZIT + IVER dose, each treated volunteer will be followed for 1 hour to observe the appearance of any side effects, then a breakfast will be offered. Head lice and nits will be searched on D1, D7, D15 and D28 for each volunteer and the hair taken on D2, D5, D7, D15 and D28. Possibly, before each treatment, Stool samples will be taken systematically on day 1 and after treatment on day 15 at any participant infested with head lice to identify intestinal parasites (load parasite in helminthiasis) to evaluate also the efficacy of ivermectin on these parasites. Sociodemographic, clinical, dose and type of material taken biological will be documented. Data on co-infections (body lice, Sarcoptes scabeii) will also be collected and reported on the study register. Each volunteer will have an identification number (ID). Only, the principal investigator, the coordinator and the investigators can access sensitive information if they exist. Data will be entered immediately by a data entry agent. The investigators will sleep on the sites and will face possible cases of effects undesirable. Regular visits will be scheduled on D2, D5, D7, D15 and D28. A clinical monitor will stay with the team on the field of D2, D5, D7, D15 and D28. A Clinical Research Organisation (CRO) will ensure the external monitoring of the study (1 site initiation visit, 2 monitoring visits and 1 visit closing of the test). It will also be scheduled for a visit by Comité National d'Ethique en Santé (CNERS) members on the field according to their schedule. All willing participants and completing the eligibility criteria for entry into this study, will be taken on a single treatment arm Azithromycin-Ivermectin in orodispersible tablets. The evaluation of the answer therapy will be done on D7 and / or D15.

ELIGIBILITY:
Includes lists of Inclusion Criteria:

* body weight ≥ 15 kg for oral administration to ivermectin, • Obtain the signed informed consent of the parent or caregiver for his participation in the study.

Includes lists of Criteria Exclusion:

* Refusal of participation,

  * Non-residents in the villages during the study period,
  * body weight <15 kg not eligible for oral administration with ivermectin,
  * Pregnant women, who in the context of the daily medical and epidemiological monitoring of the population of Dielmo-like that of Ndiop- are identified and very early at the looking at the first signs of conception in a pregnant woman from her state of pregnancy on the basis of a proven test. In addition, before any treatment with ivermectin, will be systematically requested from each of the target women of reproductive age if she is pregnant
  * Women breastfeeding at the time of the study,

Min Age: 6 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Children, adolescents and adults infested with head lice and / or co-infestation head lice and body lice
Enrollment: 450 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-24 (Actual)

PRIMARY OUTCOMES:
Parasiticidal efficacy: disappearance of head lice (zero lice) on day 7 | Day 7
  Evaluating the efficacy of the treatment of combination of two usual drugs from volunteer subjects infested with head lice.
  To study the therapeutic efficacy of the combination Azithromycin-Ivermectin administered orally in the treatment of head lice infestations (in case of persistence of lice at D7 a second oral administration of the combination azithromycin-Ivermectin will be considered).

CONTACTS AND LOCATIONS:
Overall Officials: Cheikh Sokhna, PhD, Study Director — Institut de Recherche pour le Developpement
Locations (1):
- Institut de Recherche pour le Developpement, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided
oral communications and publications